CLINICAL TRIAL: NCT03621046
Title: A Placebo Controlled Double Blind Randomised Controlled Proof of Concept Study of Zolpidem for the Treatment of Motor and Cognitive Deficits in Late-stage Parkinson's
Brief Title: Use of Low-dose Zolpidem in Parkinson's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aston University (Other)
Collaborators: University Hospital Birmingham NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RRK6212
Record Dates: First submitted 2018-06-06; First posted 2018-08-08 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Parkinson Disease
Keywords: motor;; cognition
MeSH Terms: conditions — Parkinson Disease | interventions — Zolpidem

STUDY DESIGN:
Intervention Model Description: A placebo controlled double-blinded proof-of-concept study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Zolpidem (Experimental): A single oral zolpidem tablet (5 mg) administered in clinic and then each day for the following 3 days
  Interventions: Drug: Zolpidem
- Placebo (Placebo Comparator): A single oral placebo administered in clinic and then each day for the following 3 days
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Zolpidem — Zolpidem is a non-benzodiazepine sedative/hypnotic agent usually prescribed for insomnia.
  Other Names: Stilnoct
  Arms: Zolpidem
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study will evaluate the motor and cognitive benefits of low-dose zolpidem in Parkinson's.

DETAILED DESCRIPTION:
Zolpidem is a hypnotic drug which at sub-sedative doses has been shown to improve both motor and cognitive deficits in stroke, dementia and Parkinson's. This has led to the hypothesis that low-dose zolpidem will be effective in early-stage Parkinson's, delaying the need for dopamine-replacement interventions, as an adjunct therapy, and in late-stage Parkinson's where current interventions are ineffective for motor and cognitive decline. At present, the symptoms of late-stage Parkinson's are the most debilitating and the least well-controlled. Here, the investigators propose a placebo controlled double-blinded proof-of-concept study in order to determine the benefits of taking low-dose zolpidem in late-stage Parkinson's. The study will take place over 12 months. 28 participants, diagnosed with Parkinson's for at least 5 years will be recruited; 14 participants will take zolpidem (5 mg) and 14 placebo, each morning for 4 days. In the clinic (day 1) clinical assessments will include the motor III of the Unified Parkinson's Disease Rating Scale (UPDRS) and cognitive verbal fluency tasks which will be conducted at baseline and 1 hour following drug administration. Each participant will then be issued with a smartphone with application to objectively test their motor performance 4 times a day, over the next six days (3 days on drug, 3 days off drug). This study will provide the necessary data on drug efficacy in order to design a phase II clinical trial for the use of low-dose zolpidem in late-stage Parkinson's.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of idiopathic Parkinson's and Hoehn and Yahr score of 2.5 or more; Willing to participate and refrain from driving whist taking zolpidem/placebo; Within age range 40 to 80 years.

Exclusion Criteria:

Any contraindications as stated in Summary of Product Characteristics (SmPC) for zolpidem:- Hypersensitivity to zolpidem tartrate; Obstructive sleep apnoea; Myasthenia gravis; Severe hepatic insufficiency; Acute and/or severe respiratory depression; Psychotic illness.

and in addition: - Unable or unwilling to give informed consent ; Current therapy with central nervous system (CNS) depressants; Current therapy with Cytochrome P450 (CPY450) inhibitors or inducers (specifically CYP3A4); Pregnancy and breast feeding women; History of alcohol or substance abuse; Employed in a role that involves driving or operating heavy machinery; Participation in another interventional clinical trial.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-01-24 (Actual)

PRIMARY OUTCOMES:
Changes in motor function | 1 day
  In the clinic (day 1), motor function will be assessed before and after active/placebo administration using the Unified Parkinson's Disease Rating Scale (Part III). This involves 26 assessments (scored 0-4) including of tremor, rigidity, agility and posture. Scores therefore range from 0 to 104, the higher the score indicating reduced motor function.

SECONDARY OUTCOMES:
Changes in cognitive function | 1 day
  In the clinic (day 1), cognitive function as measured by phonetic/letter fluency and semantic/category naming tasks. These test will be conducted on day 1 before and after active / placebo administration.
  The letter fluency test involves the participant giving as many different words as possible beginning with a specific letter, in 60 seconds. The category naming tasks involves the participant giving as many different examples from a given specific category (i.e, animals) in 60 seconds. The higher the score the greater the cognitive ability.
Motor performance | 6 days
  Objective measures of motor performance will be conducted using a mobile phone application specifically designed for Parkinson's patients (see Arora et al., 2015. Parkinson's and Related Disorders 21; 650-653) which measures motor performance including: testing of posture; gait; tremor; and reaction times. The testing protocol is for all patients (active and placebo) to perform tests 4 times per day on each of days 2 - 7, 3 days while taking drug/placebo, then 3 days not taking drug/placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Ian M Stanford, BSc, PhD, Study Director — Aston University
Locations (1):
- University Hospitals Birmingham NHS Foundation Trust, Birmingham, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided